CLINICAL TRIAL: NCT01726114
Title: A Clinical Study to Evaluate the Performance of the C8 MediSensors Optical Glucose Monitor™ During On-Site Testing and Real Time Use Monitoring
Brief Title: A Clinical Study of the C8 MediSensors Optical Glucose Monitor™
Acronym: Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C8 MediSensors, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: C8CSP_19042012
Record Dates: First submitted 2012-10-31; First posted 2012-11-14 (Estimated); Last update posted 2013-03-26 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Diabetes Mellitus; continuous Glucose Monitor
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Non-invasive Optical Glucose Monitor™ (Experimental): Test device
  Interventions: Device: Non-invasive Optical Glucose Monitor™; Device: YSI blood glucose analyzer

INTERVENTIONS:
Device: Non-invasive Optical Glucose Monitor™ — Test device
  Other Names: Continuous glucose monitor
Device: YSI blood glucose analyzer — Reference device
  Other Names: Yellow Springs Instruments (YSI) blod glucose analyzer

SUMMARY:
The purpose of this study is to compare glucose measurements from the C8 MediSensors non-invasive Optical Glucose Monitor™ System to blood glucose measurements from the Yellow Springs Instrument(YSI) blood glucose analyzer.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, open label study to evaluate the performance of the C8 MediSensors non-invasive Optical Glucose Monitor™ on individuals with diabetes mellitus. Capillary blood samples will be obtained throughout a daily study session; the study session may last for up to 12 hours. Blood glucose will be measured on a YSI blood glucose analyzer. Subjects may adjust food intake and insulin administration so device performance is evaluated across a broad range of glucose concentrations. Glucose measurements will be time matched and paired for comparison. Skin effects and adverse events will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Understands and agrees to comply with study instructions.
3. Read, understood, signed and dated the Informed Consent Form.

Exclusion Criteria:

1. Pregnancy.
2. Extensive skin changes or diseases that preclude wearing the test device at the proposed wear site(s) (e.g., extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis).
3. Employed by a company within the diabetes field other than the study sponsor.
4. Medical history or any condition that may, in the opinion of the investigator, compromise the subject's ability to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Performance of the test device in comparison to the reference device | 6 months
  The primary objective is to characterize the accuracy of the non-invasive glucose measurements from the Optical Glucose Monitor™ to blood glucose measurements on a sample size of approximately 30 subjects with 1000 time matched, paired data points.

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clincal, Regulatory, Quality, Principal Investigator — C8 MediSensors, Inc.
Locations (1):
- C8 MediSensors, Inc., San Jose, California, United States